CLINICAL TRIAL: NCT01984892
Title: Treatment of Solid Tumors With Intratumoral Hiltonol® (Poly-ICLC): A Phase II Clinical Study
Brief Title: Treatment of Solid Tumors With Intratumoral Hiltonol® (Poly-ICLC)
Acronym: Hiltonol
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI discretion, low enrollment
Sponsor: Nina Bhardwaj (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nina Bhardwaj, Director, Immunotherapy Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1687; BB-43984 (Other Grant/Funding Number: Mount Sinai School of Medicine - Departmental Funds)
Record Dates: First submitted 2013-11-05; First posted 2013-11-15 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Melanoma; Squamous Cell Carcinoma of the Head and Neck; Squamous Cell Carcinoma of the Skin; Sarcoma of the Skin; Basal Cell Cancer of the Skin; Breast Cancer
Keywords: Autologous Vaccination; Intratumoral Injections; Intramuscular Injections; Advanced Accessible Solid Tumors; Poly-ICLC; Phase II Clinical Trial; Safety; Efficacy; Autovaccination; In Situ; Host Targeted Strategy; Overall Survival; Immunotherapy; Adjuvant
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms | interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IT and IM injections Poly-ICLC (Experimental): Enrolled patients will receive two cycles of Poly-ICLC treatment. Each priming (intratumoral injections - IT) and boosting (intramuscular injections - IM) treatment course will constitute one cycle.
  Interventions: Drug: Poly-ICLC

INTERVENTIONS:
Drug: Poly-ICLC — Cycle 1-Weeks 1 and 2: 1mg Poly-ICLC intratumoral (IT) injections (t=6) into same lesion over 2 weeks.
  Weeks 3-9: 1mg Poly-ICLC 2x/week intramuscularly (IM) into thighs or upper arms.
  Week 10: No treatment. CT scan of chest, abdomen, pelvis and extremities or neck; possible MRI brain scan.
  Cycle 2-Weeks 11 and 12: 1mg Poly-ICLC IT injections (t=6) into same lesion over 2 weeks.
  Weeks 13-19 - 1mg Poly-ICLC 2x/weekly IM in thighs or upper arms.
  Weeks 20-26: no treatment. Week 26, evaluate response in absence of inflammation.
  Maintenance - Weeks 27-36: For patients with stable disease or response; IM poly-ICLC injections; evaluation of clinical and immune response. Week 38 repeat tumor assessment, optional biopsy
  Follow Up via phone every 3 months for 30months, after completion of treatments.
  Other Names: Hiltonol®

SUMMARY:
The purpose of this study is to test the safety of a course of injections containing Poly-ICLC in patients with advanced solid tumors that can be easily and safely reached with a needle.

Poly-ICLC is a compound that has been used to help the body in its fight against cancer.

DETAILED DESCRIPTION:
We hypothesize that this therapeutic in-situ autovaccination strategy is comprised of three immunomodulatory steps. The first is the innate immune local tumor killing induced by intratumoral Hiltonol (via NK, TNF, etc). A very close second step is optimal Th1-weighted priming through the in-situ combination of the poly-ICLC danger signal with the tumor antigens released in step 1 and further processed and cross-presented by poly-ICLC activated mDC, etc. The repeated administration of the Hiltonol danger signal IT in the context of the patient's own tumor antigens and in a way that mimics a natural viral infection may be critical to this step. Once the system is optimally primed, the third step is targeting and maintenance of the immune response and its facilitation at remote tumor sites with IM poly-ICLC through chemokine release, inflammasome activation and other costimulatory factors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma, squamous head and neck cancer, sarcoma, squamous cell carcinoma of the skin, basal cell skin cancer, or breast cancer
* Sarcoma Patients must be @ least14 yrs of age; all others 18 yrs of age or older.
* Un-resectable disease. Patients with resectable disease may be enrolled after having refused surgery and documented consultation with a surgeon.
* Disease progressed through @ least 1 systemic therapy or through local irradiation within the preceding 6 mos.
* Radiologically or visually measurable recurrent or metastatic disease and @ least 10mm in longest dimension.
* At least 1 accessible primary or metastatic tumor site that can be readily injected IT with poly-ICLC with or without ultrasound guidance. Lesion can be superficial cutaneous, subcutaneous or within a readily accessible lymph node & must measure @ least 10mm in longest dimension.
* Tumor site injection cannot have been irradiated within 8 wks of C1D1
* ECOG performance status ≤ 2.
* Normal hematologic, renal & liver function. INR<2 if off of anticoagulation. Patients on anticoagulation therapy with an INR>2 may be enrolled at the discretion of the investigator.
* Patients able to provide informed consent.
* Must agree to follow acceptable birth control methods and continue for @ least 2 mos. after last poly-ICLC dose. Women of childbearing potential must have a (-) pregnancy test.

Exclusion Criteria:

* Serious concurrent infection or medical illness.
* Bulky intracranial metastatic disease with shift of midline structures or progressive brain metastasis. Administration of immunotherapy or conventional chemotherapy treatments for metastatic cancer within 4 wks of C1D1
* Radiation treatments within 4 wks of C1D1
* AIDS defined as a CD4 count < then 200 in the context of HIV sero-positivity or chronically is taking immunosuppressive medication such as steroids or transplant related medications.
* Life expectancy of < than 6 mos.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Brody JD, Ai WZ, Czerwinski DK, Torchia JA, Levy M, Advani RH, Kim YH, Hoppe RT, Knox SJ, Shin LK, Wapnir I, Tibshirani RJ, Levy R. In situ vaccination with a TLR9 agonist induces systemic lymphoma regression: a phase I/II study. J Clin Oncol. 2010 Oct 1;28(28):4324-32. doi: 10.1200/JCO.2010.28.9793. Epub 2010 Aug 9. PMID 20697067
- [Background] Nathanson JA, Greengard P. "Second messengers" in the brain. Sci Am. 1977 Aug;237(2):109-19. No abstract available. PMID 18797
- [Background] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672
- [Background] Cella M, Salio M, Sakakibara Y, Langen H, Julkunen I, Lanzavecchia A. Maturation, activation, and protection of dendritic cells induced by double-stranded RNA. J Exp Med. 1999 Mar 1;189(5):821-9. doi: 10.1084/jem.189.5.821. PMID 10049946
- [Background] Chew V, Tow C, Huang C, Bard-Chapeau E, Copeland NG, Jenkins NA, Weber A, Lim KH, Toh HC, Heikenwalder M, Ng IO, Nardin A, Abastado JP. Toll-like receptor 3 expressing tumor parenchyma and infiltrating natural killer cells in hepatocellular carcinoma patients. J Natl Cancer Inst. 2012 Dec 5;104(23):1796-807. doi: 10.1093/jnci/djs436. Epub 2012 Nov 29. PMID 23197495
- [Background] Cho HI, Lee YR, Celis E. Interferon gamma limits the effectiveness of melanoma peptide vaccines. Blood. 2011 Jan 6;117(1):135-44. doi: 10.1182/blood-2010-08-298117. Epub 2010 Oct 1. PMID 20889921
- [Background] Davies ME, Field AK. Effect of poly I:C/poly-L-lysine (poly ICL) on the development of murine osteogenic sarcoma. J Interferon Res. 1983;3(1):89-95. doi: 10.1089/jir.1983.3.89. PMID 6573430
- [Background] Flynn BJ, Kastenmuller K, Wille-Reece U, Tomaras GD, Alam M, Lindsay RW, Salazar AM, Perdiguero B, Gomez CE, Wagner R, Esteban M, Park CG, Trumpfheller C, Keler T, Pantaleo G, Steinman RM, Seder R. Immunization with HIV Gag targeted to dendritic cells followed by recombinant New York vaccinia virus induces robust T-cell immunity in nonhuman primates. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):7131-6. doi: 10.1073/pnas.1103869108. Epub 2011 Apr 5. PMID 21467219
- [Background] Geiss G, Jin G, Guo J, Bumgarner R, Katze MG, Sen GC. A comprehensive view of regulation of gene expression by double-stranded RNA-mediated cell signaling. J Biol Chem. 2001 Aug 10;276(32):30178-82. doi: 10.1074/jbc.c100137200. PMID 11487589
- [Background] Hoos A, Eggermont AM, Janetzki S, Hodi FS, Ibrahim R, Anderson A, Humphrey R, Blumenstein B, Old L, Wolchok J. Improved endpoints for cancer immunotherapy trials. J Natl Cancer Inst. 2010 Sep 22;102(18):1388-97. doi: 10.1093/jnci/djq310. Epub 2010 Sep 8. PMID 20826737
- [Background] Houot R, Levy R. T-cell modulation combined with intratumoral CpG cures lymphoma in a mouse model without the need for chemotherapy. Blood. 2009 Apr 9;113(15):3546-52. doi: 10.1182/blood-2008-07-170274. Epub 2008 Oct 21. PMID 18941113
- [Background] Huang CC, Duffy KE, San Mateo LR, Amegadzie BY, Sarisky RT, Mbow ML. A pathway analysis of poly(I:C)-induced global gene expression change in human peripheral blood mononuclear cells. Physiol Genomics. 2006 Jul 12;26(2):125-33. doi: 10.1152/physiolgenomics.00002.2006. Epub 2006 Mar 22. PMID 16554548
- [Background] Kajiwara K, Morishima H, Akiyama K, Yanagihara Y. Expression and function of the inducible costimulator ligand B7-H2 in human airway smooth muscle cells. Allergol Int. 2009 Dec;58(4):573-83. doi: 10.2332/allergolint.09-OA-0113. Epub 2009 Sep 25. PMID 19776675
- [Background] Longhi MP, Trumpfheller C, Idoyaga J, Caskey M, Matos I, Kluger C, Salazar AM, Colonna M, Steinman RM. Dendritic cells require a systemic type I interferon response to mature and induce CD4+ Th1 immunity with poly IC as adjuvant. J Exp Med. 2009 Jul 6;206(7):1589-602. doi: 10.1084/jem.20090247. Epub 2009 Jun 29. PMID 19564349
- [Background] Lu B, Nakamura T, Inouye K, Li J, Tang Y, Lundback P, Valdes-Ferrer SI, Olofsson PS, Kalb T, Roth J, Zou Y, Erlandsson-Harris H, Yang H, Ting JP, Wang H, Andersson U, Antoine DJ, Chavan SS, Hotamisligil GS, Tracey KJ. Novel role of PKR in inflammasome activation and HMGB1 release. Nature. 2012 Aug 30;488(7413):670-4. doi: 10.1038/nature11290. PMID 22801494
- [Background] Maluish AE, Reid JW, Crisp EA, Overton WR, Levy H, Foon KA, Herberman RB. Immunomodulatory effects of poly(I,C)-LC in cancer patients. J Biol Response Mod. 1985 Dec;4(6):656-63. PMID 4087034
- [Background] Gbewonyo WS, Candy DJ. Separation of insecticidal components from an extract of the roots of male Piper guineense (west African black pepper) by gas chromatography. Toxicon. 1992 Sep;30(9):1037-42. doi: 10.1016/0041-0101(92)90048-a. PMID 1440640
- [Background] Mitsuhashi M. Ex vivo simulation of leukocyte function: stimulation of specific subset of leukocytes in whole blood followed by the measurement of function-associated mRNAs. J Immunol Methods. 2010 Dec 15;363(1):95-100. doi: 10.1016/j.jim.2010.10.002. Epub 2010 Oct 15. PMID 20951704
- [Background] Morgan ET, Norman CA. Pretranslational suppression of cytochrome P-450h (IIC11) gene expression in rat liver after administration of interferon inducers. Drug Metab Dispos. 1990 Sep-Oct;18(5):649-53. PMID 1706245
- [Background] Nierkens S, den Brok MH, Sutmuller RP, Grauer OM, Bennink E, Morgan ME, Figdor CG, Ruers TJ, Adema GJ. In vivo colocalization of antigen and CpG [corrected] within dendritic cells is associated with the efficacy of cancer immunotherapy. Cancer Res. 2008 Jul 1;68(13):5390-6. doi: 10.1158/0008-5472.CAN-07-6023. PMID 18593941
- [Background] North RJ, Dunn PL, Havell EA. A role for tumor necrosis factor in poly(I:C)-induced hemorrhagic necrosis and T-cell-dependent regression of a murine sarcoma. J Interferon Res. 1991 Dec;11(6):333-40. doi: 10.1089/jir.1991.11.333. PMID 1839310
- [Background] Pedrazzoli P, Secondino S, Perfetti V, Comoli P, Montagna D. Immunotherapeutic Intervention against Sarcomas. J Cancer. 2011;2:350-6. doi: 10.7150/jca.2.350. Epub 2011 Jun 13. PMID 21716856
- [Background] Pilaro AM, Taub DD, McCormick KL, Williams HM, Sayers TJ, Fogler WE, Wiltrout RH. TNF-alpha is a principal cytokine involved in the recruitment of NK cells to liver parenchyma. J Immunol. 1994 Jul 1;153(1):333-42. PMID 8207246
- [Background] Rosenfeld MR, Chamberlain MC, Grossman SA, Peereboom DM, Lesser GJ, Batchelor TT, Desideri S, Salazar AM, Ye X. A multi-institution phase II study of poly-ICLC and radiotherapy with concurrent and adjuvant temozolomide in adults with newly diagnosed glioblastoma. Neuro Oncol. 2010 Oct;12(10):1071-7. doi: 10.1093/neuonc/noq071. Epub 2010 Jul 8. PMID 20615924
- [Background] Salazar AM, Levy HB, Ondra S, Kende M, Scherokman B, Brown D, Mena H, Martin N, Schwab K, Donovan D, Dougherty D, Pulliam M, Ippolito M, Graves M, Brown H, Ommaya A. Long-term treatment of malignant gliomas with intramuscularly administered polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose: an open pilot study. Neurosurgery. 1996 Jun;38(6):1096-103; discussion 1103-4. PMID 8727138
- [Background] Salem ML, El-Naggar SA, Kadima A, Gillanders WE, Cole DJ. The adjuvant effects of the toll-like receptor 3 ligand polyinosinic-cytidylic acid poly (I:C) on antigen-specific CD8+ T cell responses are partially dependent on NK cells with the induction of a beneficial cytokine milieu. Vaccine. 2006 Jun 12;24(24):5119-32. doi: 10.1016/j.vaccine.2006.04.010. Epub 2006 May 2. PMID 16704888
- [Background] Sivori S, Falco M, Della Chiesa M, Carlomagno S, Vitale M, Moretta L, Moretta A. CpG and double-stranded RNA trigger human NK cells by Toll-like receptors: induction of cytokine release and cytotoxicity against tumors and dendritic cells. Proc Natl Acad Sci U S A. 2004 Jul 6;101(27):10116-21. doi: 10.1073/pnas.0403744101. Epub 2004 Jun 24. PMID 15218108
- [Background] Stahl-Hennig C, Eisenblatter M, Jasny E, Rzehak T, Tenner-Racz K, Trumpfheller C, Salazar AM, Uberla K, Nieto K, Kleinschmidt J, Schulte R, Gissmann L, Muller M, Sacher A, Racz P, Steinman RM, Uguccioni M, Ignatius R. Synthetic double-stranded RNAs are adjuvants for the induction of T helper 1 and humoral immune responses to human papillomavirus in rhesus macaques. PLoS Pathog. 2009 Apr;5(4):e1000373. doi: 10.1371/journal.ppat.1000373. Epub 2009 Apr 10. PMID 19360120
- [Background] Wick DA, Webb JR. A novel, broad spectrum therapeutic HPV vaccine targeting the E7 proteins of HPV16, 18, 31, 45 and 52 that elicits potent E7-specific CD8T cell immunity and regression of large, established, E7-expressing TC-1 tumors. Vaccine. 2011 Oct 13;29(44):7857-66. doi: 10.1016/j.vaccine.2011.07.090. Epub 2011 Aug 2. PMID 21816200
- [Background] Wong JP, Christopher ME, Viswanathan S, Dai X, Salazar AM, Sun LQ, Wang M. Antiviral role of toll-like receptor-3 agonists against seasonal and avian influenza viruses. Curr Pharm Des. 2009;15(11):1269-74. doi: 10.2174/138161209787846775. PMID 19355966
- [Background] Zhu X, Fallert-Junecko BA, Fujita M, Ueda R, Kohanbash G, Kastenhuber ER, McDonald HA, Liu Y, Kalinski P, Reinhart TA, Salazar AM, Okada H. Poly-ICLC promotes the infiltration of effector T cells into intracranial gliomas via induction of CXCL10 in IFN-alpha and IFN-gamma dependent manners. Cancer Immunol Immunother. 2010 Sep;59(9):1401-9. doi: 10.1007/s00262-010-0876-3. Epub 2010 Jun 12. PMID 20549206
- [Background] Zhu X, Nishimura F, Sasaki K, Fujita M, Dusak JE, Eguchi J, Fellows-Mayle W, Storkus WJ, Walker PR, Salazar AM, Okada H. Toll like receptor-3 ligand poly-ICLC promotes the efficacy of peripheral vaccinations with tumor antigen-derived peptide epitopes in murine CNS tumor models. J Transl Med. 2007 Feb 12;5:10. doi: 10.1186/1479-5876-5-10. PMID 17295916
- [Background] van der Most RG, Currie A, Robinson BW, Lake RA. Cranking the immunologic engine with chemotherapy: using context to drive tumor antigen cross-presentation towards useful antitumor immunity. Cancer Res. 2006 Jan 15;66(2):601-4. doi: 10.1158/0008-5472.CAN-05-2967. PMID 16423984
- [Derived] Salazar AM, Erlich RB, Mark A, Bhardwaj N, Herberman RB. Therapeutic in situ autovaccination against solid cancers with intratumoral poly-ICLC: case report, hypothesis, and clinical trial. Cancer Immunol Res. 2014 Aug;2(8):720-4. doi: 10.1158/2326-6066.CIR-14-0024. Epub 2014 May 6. PMID 24801836

RESULTS

PARTICIPANT FLOW:
Groups:
- IT and IM Injections Poly-ICLC: Enrolled patients received two cycles of Poly-ICLC treatment. Each priming (intratumoral injections - IT) and boosting (intramuscular injections - IM) treatment course will constitute one cycle.
  Poly-ICLC: Cycle 1-Weeks 1 and 2: 1mg Poly-ICLC intratumoral (IT) injections (t=6) into same lesion over 2 weeks.
  Weeks 3-9: 1mg Poly-ICLC 2x/week intramuscularly (IM) into thighs or upper arms.
  Week 10: No treatment. CT scan of chest, abdomen, pelvis and extremities or neck; possible MRI brain scan.
  Cycle 2-Weeks 11 and 12: 1mg Poly-ICLC IT injections (t=6) into same lesion over 2 weeks.
  Weeks 13-19 - 1mg Poly-ICLC 2x/weekly IM in thighs or upper arms. Weeks 20-26: no treatment. Week 26, evaluate response in absence of inflammation.
  Maintenance - Weeks 27-36: For patients with stable disease or response; IM poly-ICLC injections; evaluation of clinical and immune response. Week 38 repeat tumor assessment, optional biopsy
Period: Overall Study
Arm/Group | IT and IM Injections Poly-ICLC
Started | 8
Completed | 1 (1 completed all study visits up until the termination of the study, last study visit not done.)
Not Completed | 7
Not completed — Progressive disease | 7

BASELINE CHARACTERISTICS:
Groups:
- Participants With Stage 4 Cancer: Enrolled patients received two cycles of Poly-ICLC treatment. Each priming (intratumoral injections - IT) and boosting (intramuscular injections - IM) treatment course will constitute one cycle.
  Poly-ICLC: Cycle 1-Weeks 1 and 2: 1mg Poly-ICLC intratumoral (IT) injections (t=6) into same lesion over 2 weeks.
  Weeks 3-9: 1mg Poly-ICLC 2x/week intramuscularly (IM) into thighs or upper arms.
  Week 10: No treatment. CT scan of chest, abdomen, pelvis and extremities or neck; possible MRI brain scan.
  Cycle 2-Weeks 11 and 12: 1mg Poly-ICLC IT injections (t=6) into same lesion over 2 weeks.
  Weeks 13-19 - 1mg Poly-ICLC 2x/weekly IM in thighs or upper arms. Weeks 20-26: no treatment. Week 26, evaluate response in absence of inflammation.
  Maintenance - Weeks 27-36: For patients with stable disease or response; IM poly-ICLC injections; evaluation of clinical and immune response. Week 38 repeat tumor assessment, optional biopsy
Arm/Group | Participants With Stage 4 Cancer
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 70 [53 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival defined as the time in weeks from study entry until tumor progression defined using the Wolchok criteria or death. Patients who are alive and free from progression on the date of closing follow-up will be censored on that date.
  In order to minimize the potential for misdiagnosis of pseudoprogression, related to early inflammation, tumor measurement for determination of progression will be made at the earliest at 26 weeks.
Time Frame: average 52 weeks
Measure: Number; unit: weeks
Arm/Group | Participants With Stage 4 Cancer
Number analyzed (Participants) | 1
weeks | 41

2. Secondary Outcome: Therapeutic Effect in Treated Patients
Description: Induction of innate and/or an adaptive, specific anti-tumor T cell immune response in the injected tumor lesion and also systemically.
Time Frame: 24 months
Population: study terminated early, data not collected. study terminated before all study visits completed. this 24 month visit was not done.
Arm/Group | Participants With Stage 4 Cancer
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Overall Survival in Treated Patients
Description: Patients who are alive on the date of closing follow-up, or 30 months after completing all study treatments, will be censored on that date
Time Frame: up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Stage 4 Cancer
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Arm/Group | Participants With Stage 4 Cancer
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 4/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Stage 4 Cancer (N=8)
Periosteal inflammation and necrosis (Musculoskeletal and connective tissue disorders) | 1
Fatigue (General disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes